CLINICAL TRIAL: NCT03497013
Title: Effect of tDCS on Cognition, Symptoms in Chronic Schizophrenia Patients With Tardive dyskinesia_a Randomized, Double-blind, Sham-controlled Trial
Brief Title: Effect of tDCS on Cognition, Symptoms in Chronic Schizophrenia Patients With Tardive Dyskinesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suzhou Psychiatric Hospital (Other)
Responsible Party: Principal Investigator, Xiang-Dong Du, Associate Professor, Suzhou Psychiatric Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SS201752; Szzx201509 (Other Grant/Funding Number: Suzhou Key Medical Center for Psychiatric Diseases); SS201752 (Other Grant/Funding Number: Scientific and Technological Program of Suzhou)
Record Dates: First submitted 2018-04-03; First posted 2018-04-13 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Tardive Dyskinesia
Keywords: transcranial Direct Current Stimulation; Randomized Controlled Trial; Schizophrenia; Tardive Dyskinesia; Abnormal Involuntary Movements Scale; Tardive Dyskinesia Rating Scale; Cognition
MeSH Terms: conditions — Tardive Dyskinesia; Schizophrenia

STUDY DESIGN:
Intervention Model Description: The aim of the study was to evaluate the efficacy, safety, and cognitive function of transcranial direct current stimulation (tDCS) in chronic schizophrenia patients with tardive dyskinesia (TD).
Who Masked: Participant, Outcomes Assessor
Masking Description: This study is a randomized, double-blind, sham-controlled clinical trial.All patients received 2-mA anodal left/cathodal right prefrontal tDCS treatment (fifteen 30-minutes sessions: Monday to Friday once daily, every other week to do a group of treatment). All evaluations were performed at baseline, the end of 3rd weeks, 5th weeks, and 7th weeks by 2 psychiatrists blinded to the treatment assigned. Inter-rater reliability was satisfactory(ka=0.86).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Experimental): All patients received 2-mA anodal left/cathodal right prefrontal tDCS treatment (fifteen 30-minutes sessions: Monday to Friday once daily, every other week to do a group of treatment).
  Interventions: Device: Active tDCS
- Sham tDCS (Sham Comparator): For sham stimulation, the device was set to turn off after 30 seconds(study model).
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — All patients received 2-mA anodal left/cathodal right prefrontal tDCS treatment (fifteen 30-minutes sessions: Monday to Friday once daily, every other week to do a group of treatment).
  Arms: Active tDCS
Device: Sham tDCS — For sham stimulation, the device was set to turn off after 30 seconds(study model).
  Arms: Sham tDCS

SUMMARY:
The aim of the study was to evaluate the efficacy, safety, and cognitive function of transcranial direct current stimulation (tDCS) in chronic schizophrenia patients with tardive dyskinesia (TD).

DETAILED DESCRIPTION:
This study is a randomized, double-blind, sham-controlled clinical trial. 60 patients with TD were randomly allocated to active (n=30) or sham tDCS groups (n=30). All patients received 2-mA anodal left/cathodal right prefrontal tDCS treatment (fifteen 30-minutes sessions: Monday to Friday once daily, every other week to do a group of treatment). Abnormal Involuntary Movements Scale (AIMS), Tardive Dyskinesia Rating Scale (TDRS), Assessment of Negative Symptoms(SANS), the Positive and Negative symptom scale(PANSS), and the Cambridge Neuropsychological Test Automatic Battery (CANTAB) were assessed in patients. All evaluations were scored at baseline, the end of 3rd weeks, 5th weeks, and 7th weeks. Side effects of tDCS were assessed with an experimenter-administered open-ended questionnaire during the whole experiment.

ELIGIBILITY:
Inclusion Criteria:

1. Right-handed;
2. meeting the diagnosis of schizophrania;
3. had been receiving antipsychotic drugs for at least 12 months;
4. at least one AIMS item rated(moderate) or at least two AIMS items rated ≥2(mild);
5. All patients volunteered to participate in this study.

Exclusion Criteria:

1. organic disorder that could cause movement disorders, mental retardation,and a history of substance dependence(except nicotine);
2. with serious physical illness(e.g.severe cardiovascular diseases);
3. with color blindness/weakness, stuttering, deafness.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2020-08-11 (Actual); Study Completion 2020-08-11 (Actual)

PRIMARY OUTCOMES:
Abnormal Involuntary Movements Scale | Change from baseline AIMS(items1-7) total scores at 3 weeks and 5 weeks and 7 weeks
  The primary outcome measure was the severity of TD symptoms, which was measured by the AIMS total score(the sum of items 1-7).The range for subscale scores(items1-7) is between 0-28 scores and the higher values represent a worse outcome.

SECONDARY OUTCOMES:
Tardive Dyskinesia Rating Scale | Change from baseline TDRS total scores at 3 weeks and 5 weeks and 7 weeks
  The severity of TD symptoms were also measured by the total TDRS score and the orofacial dyskinesia subscale scores, trunk and limb dyskinesia subscale scores. The range for TDRS total score is between 44-264 scores and the orofacial dyskinesia subscale scores are between16-96 scores , the trunk and limb dyskinesia subscale scores are between 24-144 scores.The higher values represent a worse outcome.
Safety and Tolerabilit | We assessed the side affects during and after tDCS.
  Side effects of tDCS were assessed with an experimenter-administered open-ended questionnaire during the whole experiment. The questionnaire contained rating scales regarding the presence and severity of headache, difficulties in concentrating, acute mood changes, visual perceptual changes and any discomforting sensation like pain, tingling, itching or burning under the electrodes.
Scale for the Assessment of Negative Symptoms | Change from baseline SANS total scores at 5 weeks
  Negative symptoms were assessed with SANS. The range for SANS total scores is between 0-120 scores and the higher values represent a worse outcome.
Positive and Negative symptom scale | Change from baseline PANSS total scores at 5 weeks
  Psychopathology was measured by the total PANSS score and the positive, negative, and general psychopathology subscale scores. The range for PANSS total score is between 30-210 scores and the positive subscale scores are between 7-49 scores and the negative subscale scores are between 7-49 scores and the general psychopathology total scores are between 16-112 scores.
Cambridge Neuropsychological Test Automatic Battery | Change from baseline cognitive function at 3 weeks and 5 weeks and 7 weeks
  Each patient was given a series of computerized tests from the Cambridge Neuropsychological Test Automated Battery. The language-independent tests and touch screen technology deliver rapid and non-invasive cognitive assessment. Executive and memory function were assessed with the following three tasks:The Pattern Recognition Memory (PRM), Intra/Extradimensional Set Shift (IED), and Spatial Working Memory.

CONTACTS AND LOCATIONS:
Overall Officials: Guangzhong Yin, MD, Study Chair — Suzhou Guangji Hospital
Locations (2):
- China (2):
  - Suzhou Psychiatric Hospital, Suzhou, Jiangsu
  - Suzhou, Suzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou Y, Xia X, Zhao X, Yang R, Wu Y, Liu J, Lyu X, Li Z, Zhang G, Du X. Efficacy and safety of Transcranial Direct Current Stimulation (tDCS) on cognitive function in chronic schizophrenia with Tardive Dyskinesia (TD): a randomized, double-blind, sham-controlled, clinical trial. BMC Psychiatry. 2023 Aug 24;23(1):623. doi: 10.1186/s12888-023-05112-0. PMID 37620825

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-11): https://cdn.clinicaltrials.gov/large-docs/13/NCT03497013/Prot_SAP_000.pdf
  • Informed Consent Form (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT03497013/ICF_001.pdf